CLINICAL TRIAL: NCT06301776
Title: A Prospective, Experimental, Multicenter, Open-label, Randomized, Controlled Trial of 3-month Dual Antiplatelet Therapy Followed by Ticagrelor Versus 6-month Dual Antiplatelet Therapy Followed by Ticagrelor After Implanting Bridge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Lianbo Gao, Chief Physician, The Fourth Affiliated Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bridge-2023-02-0A
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Brain Disease; Vertebral Artery Stenosis
MeSH Terms: conditions — Brain Diseases; Vertebrobasilar Insufficiency | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 3 Months DAPT+9 months ticagrelor monotherapy after Bridge(MicroPort NeuroTech, Shanghai, China) implantation
  Interventions: Drug: Ticagrelor
- Control group (Active Comparator): 6 Months DAPT+6 months ticagrelor monotherapy after Bridge(MicroPort NeuroTech, Shanghai, China) implantation
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — To compare the safety and efficacy of different DAPT duration combined with ticagrelor monotherapy.

SUMMARY:
To compare the incidence of the composite endpoints of non-fatal ischaemic stroke, transient ischaemia (TIA) and all-cause mortality at 12-month follow-up after implantation of Bridge for the treatment of symptomatic vertebral artery stenosis in subjects who had been taking different durations of dual-antiplatelet therapy (3 vs 6 months) and ticagrelor monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are suitable for Bridge implantation
* Symptomatic vertebral artery stenosis with a history of posterior circulation-related ischaemic stroke or TIA despite the use of at least one antithrombotic medications and intervention for risk factors
* Responsible vertebral artery stenosis (≥70% stenosis, measured by the NASCET method ) confirmed by DSA imaging
* The patient and/or his/her authorised person understands the purpose of the study, agrees to participate in the study and signs the informed consent form

Exclusion Criteria:

* mRS≥3
* Presence of tandem stenotic lesions in the target lesion areaor combined basilar artery stenosis Presence of ≥2 stenotic cerebrovascular lesions requiring concurrent intervention The presence of severe tortuosity or calcification of the target vessel, or the presence of extensive abnormal vascular structural variants that are difficult for catheters or stents to pass or cannot be implanted
* Lesions or stenosis that is too large and beyond the specification of the stent
* Non-atherosclerotic stenosis such as atrial fibrillation, vasculitis stenosis, arterial entrapment, smoky disease, active phase of arteritis, or unknown cause
* Contraindication to heparin, aspirin, tegretol, clopidogrel, or other antiplatelet drugs, and those who cannot tolerate anticoagulant and antiplatelet drug therapy
* Have had intracranial haemorrhage within 3 months
* Had a myocardial infarction or large cerebral infarction within 2 weeks
* Accompanied by other intracranial disease such as aneurysm, arteriovenous malformation, intracranial tumour, intracranial infection, etc
* Presence of active bleeding or extremely dangerous risk of haemorrhage (e.g. active peptic ulcer disease, gastrointestinal lesions with bleeding risk, malignant tumours with bleeding risk, etc.)
* Severe cardiac, hepatic, splenic, pulmonary, or renal impairment, or allergy or intolerance to contrast media, rapamycin (Rapamycin) and its derivatives, cobalt-based alloys, or polylactic acid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite endpoint of non-fatal ischaemic Stroke, TIA, and all-cause mortality at 12-months. | 365±60 days

SECONDARY OUTCOMES:
Incidence of the composite endpoint of major bleeding and hemorrhagic stroke at 12-months. | 365±60 Days
Incidence of target vessel-related stroke and neurological death at 1month | 30±7 Days
Incidence of stroke and neurological death at 12 month. | 365±60 Days
Incidence of all-cause mortality at 12 month. | 365±60 days
Incidence of in-stent-stenosis at 12 month (subgroup of imaging follow-up). | 365±60 days

CONTACTS AND LOCATIONS:
Overall Officials: Lianbo Gao, Principal Investigator — the Fourth Affilicated Hospital of China Medical University
Locations (1):
- the Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning, China